CLINICAL TRIAL: NCT01376583
Title: Running From Cancer
Brief Title: Exercise Controls Tumor Cell Growth Through AMPK Activation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Inge Holm, Administrator, Rigshospitalet, Denmark
Other Study IDs: VEK-H-3-2010-141
Record Dates: First submitted 2011-06-16; First posted 2011-06-20 (Estimated); Last update posted 2013-12-02 (Estimated); Status verified 2013-11

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Exercise; Myokines; AMPK
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bloodsamples wherefrom, serum is isolated and kept at -20 degrees celsius
Oversight: Data Monitoring Committee: No

SUMMARY:
The study investigates the explanation for the positive relation found between exercise and breastcancer.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Females age 18-30
* BMI 18-25
* Regular period

Exclusion Criteria:

* Ingestions of any hormones
* Pregnancy
* Chronic inflammation
* Elite athletes

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy Danish females in the age 18-30
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bente K Pedersen, Professor, Study Director — Centre of Inflammation and Metabolism
Locations (1):
- Centre of Inflammation and Metabolism, Copenhagen, Denmark